CLINICAL TRIAL: NCT00712231
Title: To Assess the Degree of Agreement of Anterior Chamber Depth Measurements by 2 Optical Devices (Pentacam and IOLMaster) and Compare Them With Contact Ultrasound A-Scan in Phakic and Pseudophakic Eyes.
Brief Title: Limitations of Using a Sheimpflug Image-Based Device for Measuring Anterior Chamber Depth in Pseudophakic Eyes
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Shu-Wen Chang/Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Other Study IDs: FEMH97007
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: Cataract
Keywords: pseudophakic; anterior chamber depth; Pentacam
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — no specimen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- phakic eyes: the cases did not accept any intraocular surgery
- pseudophakic eyes: tht cases did not accept any intraocular surgery expect for cataract surgery

SUMMARY:
There have been numerous studies comparing various ACD measurements in phakic eyes,while researches comparing ACD in pseudophakic eyes are less extensive. With the recent popularity of presbyopia correction, measuring the ACD will facilitate differentiating pseudophakic accommodation from pseudoaccommodation. It is thus mandatory to verify the accuracy of ACD measurement of these devices since the innovation of various IOLs in the recent decade makes this task more complicated. In this study, we will assess the limitations of using Pentacam for ACD measurement in pseudophakic eyes and compare Pentacam measurement with IOLMaster and A-scan measurements.

DETAILED DESCRIPTION:
In this prospective study, ACD was measured in 90 phakic and 94 pseudophakic eyes by Pentacam, IOLMaster and A-scan. Correlations and differences between the three measurements were investigated. The accuracy in detecting the anterior lens surface in pseudophakic eyes was also assessed.Differences in ACD-Pen, ACD-IOLM, and ACD-A were analyzed using one-way analysis of variance (ANOVA). When an overall significance of P< 0.05 was obtained, pair-wise comparisons were made using Tukey's multiple comparison t tests. The association between ACD-Pen, ACD-IOLM, and ACD-A was assessed using Pearson's correlation test. The distribution of erroneous ACD-Pen measurement for the three IOLs was analyzed with the chi-square test. In all analyses, P <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Phakic group: randomized
* Pseudophakic eyes : the cases accepted cataract surgery

Exclusion Criteria:

* Previous ocular trauma or intraocular surgery other than cataract surgery;
* Contact lens use in the past two months;
* Use of medication that might affect the pupil; corneal disease or ocular infection;
* History of ocular disease, such as

  * Dry eye syndrome
  * Uveitis
  * Glaucoma
  * Ocular tumor
* Cases with any surgical complications were also excluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ninety phakic eyes were randomly selected for study from the outpatient clinic. Ninety-four pseudophakic eyes that had a standard clear cornea phacoemulsification with one of three acrylic IOLs (MA60BM, SA60AT, SN60AT) implanted into the capsular bag by the same surgeon were also studied.
Sampling Method: Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Wen Chang, Principal Investigator — Far Eastern Memorial Hospital